CLINICAL TRIAL: NCT01516489
Title: Improving Fecal Occult Blood Test Completion Rates Among Veterans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Collaborators: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven C. Marcus, PhD, Principal Investigator, Corporal Michael J. Crescenz VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01334
Record Dates: First submitted 2012-01-19; First posted 2012-01-25 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer
Keywords: screening; colon cancer; incentives; behavioral economics
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Stage 1 Control Group (No Intervention): In the FOBT kit, individuals will receive a card that asks them to complete and return their FOBT kit within 30 days.
- $5 Incentive (Experimental): In the FOBT kit, individuals will receive a card that states that if they complete and return their FOBT kit within 30 days, they will be mailed a voucher that can be exchanged for $5 at PVAMC.
  Interventions: Behavioral: Stage 1
- $10 Incentive (Experimental): In the FOBT kit, individuals will receive a card that states that if they complete and return their FOBT kit within 30 days, they will be mailed a voucher that can be exchanged for $10 at PVAMC.
  Interventions: Behavioral: Stage 1
- $20 Incentive (Experimental): In the FOBT kit, individuals will receive a card that states that if they complete and return their FOBT kit within 30 days, they will be mailed a voucher that can be exchanged for $20 at PVAMC.
  Interventions: Behavioral: Stage 1
- $5 Voucher-Based Incentive (Experimental): In the FOBT kit, individuals will receive a card that states that if they complete and return their FOBT kit within 30 days, they will be mailed a voucher that can be exchanged for $5 at PVAMC.
  Interventions: Behavioral: Stage 2
- $50 Lottery-Based Incentive (Experimental): In the FOBT kit, individuals will receive a card that states that if they complete and return their FOBT kit within 30 days, they will have a 1 in 10 chance of being mailed a voucher that can be exchanged for $50 at PVAMC.
  Interventions: Behavioral: Stage 2
- $500 Raffle-Based Incentive (Experimental): In the FOBT kit, individuals will receive a card that states that if they complete and return their FOBT kit within 30 days, they will be entered into a raffle in which 1 randomly chosen patient (out of about 100 patients) will be mailed a check in the amount of $500.
  Interventions: Behavioral: Stage 2
- Stage 2 Control Group (No Intervention): In the FOBT kit, individuals will receive a card that asks them to complete and return their FOBT kit within 30 days.

INTERVENTIONS:
Behavioral: Stage 1 — Patients who are prescribed an FOBT kit in one of the PVAMC Primary Care clinics (i.e., Module B or C) will be randomly assigned by day to one of 4 study arms. All FOBT kits will include a card with a description of the arm that the patient has been randomized to.
  Arms: $10 Incentive; $20 Incentive; $5 Incentive
Behavioral: Stage 2 — Patients who are prescribed an FOBT kit in one of the PVAMC Primary Care clinics (i.e., Module B or C) will be randomly assigned by day to one of 4 study arms. All FOBT kits will include a card with a description of the arm that the patient has been randomized to. The exact dollar amounts for the Voucher-Based Incentive, Lottery-Based Incentive, and Raffle-Based Incentive arms will be based on the results of Stage 1.
  Arms: $5 Voucher-Based Incentive; $50 Lottery-Based Incentive; $500 Raffle-Based Incentive

SUMMARY:
This is a 4-arm cluster randomized controlled trial to evaluate whether patient financial incentives directly integrated into primary care can improve fecal occult blood test (FOBT) completion rates. We will recruit primary care patients at the Philadelphia Veterans Affairs Medical Center (PVAMC) in 2 stages. In stage 1, we hypothesize that, compared to usual care, $5, $10, $20 incentives will each lead to a statistically significant increase in the rate of FOBT completion. We also hypothesize that there will be a direct dose-response relationship between the incentive amount and rates of FOBT completion. In stage 2, we hypothesize that a lottery-based incentive and a raffle-based incentive will both lead to a statistically significant increase in the rate of FOBT completion compared to a fixed payment incentive with an equivalent dollar per patient value.

ELIGIBILITY:
Inclusion Criteria:

* PVAMC outpatients who are prescribed an FOBT kit in Module B or C during the study period.

Exclusion Criteria:

* None. All PVAMC outpatients who are prescribed an FOBT kit in Module B or C during the study period will be eligible.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1549 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
FOBT completion and return | 30 days

SECONDARY OUTCOMES:
FOBT completion rate among previously non-adherent patients and FOBT kit return time by arm | 30 days
  There are 2 secondary outcomes. First, we will compare time to FOBT kit return by arm. Second, we will compare 30 day FOBT completion rates among previously non-adherent patients (i.e., individuals who had failed to complete a prescribed FOBT kit in the year prior to the start of the study) by arm.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T Kullgren, MD, MS, MPH, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center; Steven C Marcus, PhD, Study Director — Corporal Michael J. Crescenz VA Medical Center
Locations (1):
- Philadelphia Veterans Affairs Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kullgren JT, Dicks TN, Fu X, Richardson D, Tzanis GL, Tobi M, Marcus SC. Financial incentives for completion of fecal occult blood tests among veterans: a 2-stage, pragmatic, cluster, randomized, controlled trial. Ann Intern Med. 2014 Nov 18;161(10 Suppl):S35-43. doi: 10.7326/M13-3015. PMID 25402401